CLINICAL TRIAL: NCT03365011
Title: Nitrous Oxide as Treatment for Tinnitus: A Randomized Crossover Trial
Brief Title: Nitrous Oxide Treatment for Tinnitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201606104
Record Dates: First submitted 2017-05-15; First posted 2017-12-07 (Actual); Results first posted 2018-11-06 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-11

CONDITIONS: Tinnitus
Keywords: Nitrous Oxide
MeSH Terms: conditions — Tinnitus | interventions — Endothelium-Dependent Relaxing Factors; Inhalation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo was defined as 50% nitrogen and 50% oxygen for 40 minutes.
  Participants are blinded to the order of interventions administered. Participants have been informed prior to consent that one session will contain the nitrous oxide gas mixture, and the other session will contain the placebo gas mixture.
  Interventions: Drug: Placebo gas for inhalation
- Nitrous oxide (Experimental): Nitrous oxide treatment was defined as 50% nitrous oxide and 50% oxygen for 40 minutes.
  Participants are blinded to the order of interventions administered. Participants have been informed prior to consent that one session will contain the nitrous oxide gas mixture, and the other session will contain the placebo gas mixture.
  Interventions: Drug: Nitrous oxide gas for inhalation

INTERVENTIONS:
Drug: Nitrous oxide gas for inhalation — Nitrous oxide gaseous mixture (50% nitrous oxide and 50% oxygen) for 40 minutes duration under anesthesia supervision with monitoring according to standards set by the American Society of Anesthesiologists.
  Arms: Nitrous oxide
Drug: Placebo gas for inhalation — Placebo gaseous mixture (50% nitrogen and 50% oxygen) for 40 minutes duration under anesthesia supervision with monitoring according to standards set by the American Society of Anesthesiologists.
  Arms: Placebo

SUMMARY:
Tinnitus is perception of sound without the presence of an external acoustic stimulus. Approximately 50 million Americans experience chronic tinnitus and of these, 10 million have bothersome tinnitus. The tinnitus research literature suggests that NMDA receptor antagonists may prove to be useful in reducing tinnitus. Nitrous oxide, a member of the NMDA receptor antagonist class, is a widely-used general anesthetic and sedative with a proven safety profile. The investigators hypothesized that the administration of nitrous oxide, an NMDA receptor antagonist, may be effective in treatment of tinnitus. The study design was a randomized placebo-controlled crossover trial.

DETAILED DESCRIPTION:
Subjective, idiopathic, non-pulsatile tinnitus ("tinnitus") is perception of sound without the presence of an external acoustic stimulus. Approximately 50 million Americans experience chronic tinnitus and of these, 10 million have bothersome tinnitus. Bothersome tinnitus is associated with poorer working memory, slower processing speeds and reaction times, and deficiencies in selective attention.

Currently, effective therapies for tinnitus remain limited. Examples of therapies include external sound therapy to mask the perceived sound, behavioral therapy to habituate the patient to the perceived sound, and counseling such as cognitive behavioral therapy to address the bother and impact that tinnitus has on people's lives. Surgical treatment such as nerve transection remains controversial given its lack of efficacy and adverse event profile. There are no drugs approved by the FDA for the treatment of tinnitus. Antidepressant and antianxiety medications are prescribed to patients with tinnitus with limited benefit.

Nitrous oxide is an N-methyl-D-aspartate (NMDA) receptor antagonist, a class of drugs shown to have antidepressant effects. A previous trial examined the use of nitrous oxide as a treatment for major depressive disorder (MDD). Generally, NMDA receptors promote excitation at synapses throughout the auditory pathway and play diverse roles in synaptic development and auditory information processing. In the setting of chronic damage to the auditory system, overactivation of NMDA receptors leads to aberrant spontaneous neuronal firing in the cochlea and auditory brainstem structures, which can further perpetuate damage and disease in a feed-forward mechanism. Studies by Guitton et al. and Puel et al. showed that administration of NMDA receptor antagonists prior to the administration of salicylate was effective in preventing acute excitotoxic tinnitus, establishing that salicylate induces tinnitus through its action on NMDA receptors. Thus, NMDA receptors are thought to be implicated in the generation and perpetuation of several auditory diseases including tinnitus. The investigators hypothesized that the administration of nitrous oxide, an NMDA receptor antagonist, may be a therapeutic strategy in the treatment of tinnitus.

The study was a randomized placebo-controlled crossover trial. Each participant attended two intervention sessions, one "treatment" and one "placebo". Participants eligible to participate in the study were randomly assigned to receive either placebo followed by nitrous oxide or nitrous oxide followed by placebo, according to a computer-generated randomization sequence. Only the statistician and the anesthesiology team directly involved in administration of nitrous oxide and placebo had access to the group assignments. All participants and other study team members administering survey assessments remained blinded. The two intervention sessions were held at least two weeks apart and were indistinguishable in setting, setup, and monitoring in order to maintain blinding for the participants and study team members. All intervention sessions were performed at the Washington University Clinical Research Unit, a component of the Center for Applied Research Sciences.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women 18-65 years of age
* Subjective, unilateral or bilateral, non-pulsatile tinnitus scoring "Bothered more than a little but not a lot", "Bothered a lot", or "Extremely bothered" on the Global Bothersome scale
* Able to give informed consent
* Must be able to read, write, and understand English

Exclusion Criteria:

* Bipolar disorder
* Schizophrenia
* Schizoaffective disorder
* Substance abuse or dependence (except for remote substance abuse or dependence with remission at least 1 year prior to the study and except for nicotine use disorders)
* Acute medical illness that may pose subject at risk during nitrous oxide administration
* Active psychotic symptoms
* Patients with significant pulmonary disease and/or requiring supplemental oxygen
* Contraindication against the use of nitrous oxide:
* Pneumothorax
* Bowel obstruction
* Middle ear occlusion
* Elevated intracranial pressure
* Chronic cobalamin and/or folate deficiency treated with folic acid or vitamin B12
* Pregnant patients
* Breastfeeding women
* Previous administration of NMDA-receptor antagonists (e.g., ketamine) within the last 3 months
* Tinnitus related to cochlear implantation, retrocochlear lesion, Meniere's Disease, or other known anatomic lesions of the ear or temporal bone
* Tinnitus related to a Workman's Compensation claim or litigation-related event that is still pending.
* Any medical condition, which, in the opinion of the PI, confounds study results or places the subject at greater risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shargorodsky J, Curhan GC, Farwell WR. Prevalence and characteristics of tinnitus among US adults. Am J Med. 2010 Aug;123(8):711-8. doi: 10.1016/j.amjmed.2010.02.015. PMID 20670725
- [Background] Pierce KJ, Kallogjeri D, Piccirillo JF, Garcia KS, Nicklaus JE, Burton H. Effects of severe bothersome tinnitus on cognitive function measured with standardized tests. J Clin Exp Neuropsychol. 2012;34(2):126-34. doi: 10.1080/13803395.2011.623120. Epub 2011 Dec 14. PMID 22168528
- [Background] Tunkel DE, Bauer CA, Sun GH, Rosenfeld RM, Chandrasekhar SS, Cunningham ER Jr, Archer SM, Blakley BW, Carter JM, Granieri EC, Henry JA, Hollingsworth D, Khan FA, Mitchell S, Monfared A, Newman CW, Omole FS, Phillips CD, Robinson SK, Taw MB, Tyler RS, Waguespack R, Whamond EJ. Clinical practice guideline: tinnitus. Otolaryngol Head Neck Surg. 2014 Oct;151(2 Suppl):S1-S40. doi: 10.1177/0194599814545325. PMID 25273878
- [Background] Langguth B, Elgoyhen AB. Current pharmacological treatments for tinnitus. Expert Opin Pharmacother. 2012 Dec;13(17):2495-509. doi: 10.1517/14656566.2012.739608. Epub 2012 Nov 4. PMID 23121658
- [Background] Beebe Palumbo D, Joos K, De Ridder D, Vanneste S. The Management and Outcomes of Pharmacological Treatments for Tinnitus. Curr Neuropharmacol. 2015;13(5):692-700. doi: 10.2174/1570159x13666150415002743. PMID 26467416
- [Background] Jevtovic-Todorovic V, Todorovic SM, Mennerick S, Powell S, Dikranian K, Benshoff N, Zorumski CF, Olney JW. Nitrous oxide (laughing gas) is an NMDA antagonist, neuroprotectant and neurotoxin. Nat Med. 1998 Apr;4(4):460-3. doi: 10.1038/nm0498-460. PMID 9546794
- [Background] Nagele P, Duma A, Kopec M, Gebara MA, Parsoei A, Walker M, Janski A, Panagopoulos VN, Cristancho P, Miller JP, Zorumski CF, Conway CR. Nitrous Oxide for Treatment-Resistant Major Depression: A Proof-of-Concept Trial. Biol Psychiatry. 2015 Jul 1;78(1):10-18. doi: 10.1016/j.biopsych.2014.11.016. Epub 2014 Dec 9. PMID 25577164
- [Background] Sanchez JT, Ghelani S, Otto-Meyer S. From development to disease: diverse functions of NMDA-type glutamate receptors in the lower auditory pathway. Neuroscience. 2015 Jan 29;285:248-59. doi: 10.1016/j.neuroscience.2014.11.027. Epub 2014 Nov 25. PMID 25463512
- [Background] Kaltenbach JA, Zhang J, Finlayson P. Tinnitus as a plastic phenomenon and its possible neural underpinnings in the dorsal cochlear nucleus. Hear Res. 2005 Aug;206(1-2):200-26. doi: 10.1016/j.heares.2005.02.013. PMID 16081009
- [Background] Sahley TL, Nodar RH, Musiek FE. Endogenous dynorphins: possible role in peripheral tinnitus. Int Tinnitus J. 1999;5(2):76-91. PMID 10753426
- [Background] Nicolas-Puel C, Faulconbridge RL, Guitton M, Puel JL, Mondain M, Uziel A. Characteristics of tinnitus and etiology of associated hearing loss: a study of 123 patients. Int Tinnitus J. 2002;8(1):37-44. PMID 14763234
- [Background] Guitton MJ, Dudai Y. Blockade of cochlear NMDA receptors prevents long-term tinnitus during a brief consolidation window after acoustic trauma. Neural Plast. 2007;2007:80904. doi: 10.1155/2007/80904. PMID 18301716
- [Background] Puel JL. Cochlear NMDA receptor blockade prevents salicylate-induced tinnitus. B-ENT. 2007;3 Suppl 7:19-22. PMID 18225604
- [Background] Guitton MJ, Caston J, Ruel J, Johnson RM, Pujol R, Puel JL. Salicylate induces tinnitus through activation of cochlear NMDA receptors. J Neurosci. 2003 May 1;23(9):3944-52. doi: 10.1523/JNEUROSCI.23-09-03944.2003. PMID 12736364
- [Background] Guitton MJ. Tinnitus: pathology of synaptic plasticity at the cellular and system levels. Front Syst Neurosci. 2012 Mar 8;6:12. doi: 10.3389/fnsys.2012.00012. eCollection 2012. PMID 22408611
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Standards for Basic Anesthetic Monitoring. Committee of Origin: Standards and Practice Parameters (Approved by the ASA House of Delegates on October 21, 1986, last amended on October 20, 2010, and last affirmed on October 28, 2016) https://www.asahq.org/~/media/Sites/ASAHQ/Files/Public/Resources/standards-guidelines/standards-for-basic-anesthetic-monitoring.pdf
- [Background] Meikle MB, Henry JA, Griest SE, Stewart BJ, Abrams HB, McArdle R, Myers PJ, Newman CW, Sandridge S, Turk DC, Folmer RL, Frederick EJ, House JW, Jacobson GP, Kinney SE, Martin WH, Nagler SM, Reich GE, Searchfield G, Sweetow R, Vernon JA. The tinnitus functional index: development of a new clinical measure for chronic, intrusive tinnitus. Ear Hear. 2012 Mar-Apr;33(2):153-76. doi: 10.1097/AUD.0b013e31822f67c0. PMID 22156949
- [Background] Andersson G, Westin V. Understanding tinnitus distress: introducing the concepts of moderators and mediators. Int J Audiol. 2008 Nov;47 Suppl 2:S106-11. doi: 10.1080/14992020802301670. PMID 19012118
- [Background] Duckert LG, Rees TS. Placebo effect in tinnitus management. Otolaryngol Head Neck Surg. 1984 Dec;92(6):697-9. doi: 10.1177/019459988409200618. PMID 6440090
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Derived] Hong HY, Karadaghy O, Kallogjeri D, Brown FT, Yee B, Piccirillo JF, Nagele P. Effect of Nitrous Oxide as a Treatment for Subjective, Idiopathic, Nonpulsatile Bothersome Tinnitus: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Sep 1;144(9):781-787. doi: 10.1001/jamaoto.2018.1278. PMID 30073285

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First: Participants are randomized to receive placebo during the first session, followed by nitrous oxide during the second session.
- Nitrous Oxide First: Participants are randomized to receive nitrous oxide during the first session, followed by placebo during the second session.
Period: Overall Study
Arm/Group | Placebo First | Nitrous Oxide First
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Nitrous Oxide: Participants are randomized to receive nitrous oxide during the first session, followed by placebo during the second session.
- Total: Total of all reporting groups
Arm/Group | Placebo First | Nitrous Oxide | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (9.4) | 52.8 (11.1) | 52.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 7 | 13 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 16 | 15 | 31
  Race: Black | 1 | 2 | 3
  Race: Other | 3 | 2 | 5
  Race: Did not respond | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Tinnitus Functional Index [Median (Full Range); unit: units on a scale] — The Tinnitus Functional Index (TFI) is a 25-question survey assessing tinnitus impact on quality of life. Participants were asked to rate on a scale from 0-10 the degree of unpleasantness, cognitive interference, sleep disturbance, auditory difficulties, interference with relaxation, and emotional distress associated with their tinnitus. Subscores are summed and scaled to a score of 0-100. A score less than 25 indicates mild problems due to tinnitus and little need for intervention, while a score between 25-50 indicates significant problems due to tinnitus with potential need for intervention.
  units on a scale | 42 [6 to 82] | 40 [21 to 92] | 41 [6 to 92]
Global Bothersome Scale [Count of Participants; unit: Participants]
  Not bothered | 0 | 0 | 0
  Bothered a little, but not much | 0 | 0 | 0
  Bothered more than a little, but not a lot | 12 | 12 | 24
  Bothered a lot | 7 | 5 | 12
  Extremely bothered | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Tinnitus Functional Index (TFI) Score
Description: Change of participant-reported tinnitus symptoms 1 week after each intervention.
  The Tinnitus Functional Index (TFI) is a 25-question survey assessing tinnitus impact on quality of life. Participants were asked to rate on a scale from 0-10 the degree of unpleasantness, cognitive interference, sleep disturbance, auditory difficulties, interference with relaxation, and emotional distress associated with their tinnitus. Subscores are summed and scaled to a score of 0-100. A score less than 25 indicates mild problems due to tinnitus and little need for intervention, while a score between 25-50 indicates significant problems due to tinnitus with potential need for intervention.
  A decrease in TFI score indicates decreased bother due to tinnitus over time, a better outcome. An increase in TFI score indicates increased bother due to tinnitus over time, a worse outcome.
Time Frame: Pre-intervention and 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Placebo was defined as 50% nitrogen and 50% oxygen for 40 minutes.
- Nitrous Oxide: Nitrous oxide treatment was defined as 50% nitrous oxide and 50% oxygen for 40 minutes.
Arm/Group | Placebo | Nitrous Oxide
Number analyzed (Participants) | 39 | 38
score on a scale | -1.8 (8.8) | -2.5 (11.0)

2. Secondary Outcome: Change in Global Bothersome Scale (GBS) Score
Description: Change in participant-reported tinnitus bother after each intervention.
  Global Bothersome Scale (GBS) measured participant's self-assessment of tinnitus bother on a 5-point scale ranging from "Not bothered, 0" to "Extremely bothered, 5."
  A change of 0 indicates no change in tinnitus bother over time. A change of -1 indicates somewhat improved tinnitus bother, and a change of positive 1 indicates somewhat worsened tinnitus bother. A change of positive 2 indicates significantly worsened tinnitus bother.
Time Frame: Pre-intervention and 1 week post-intervention
Measure: Number; unit: participants
Arm/Group | Placebo | Nitrous Oxide
Number analyzed (Participants) | 39 | 38
participants
  Somewhat improved, -1 | 5 | 2
  No change, 0 | 28 | 34
  Somewhat worsened, 1 | 5 | 2
  Significantly worsened, 2 | 1 | 0

3. Secondary Outcome: Patients' Global Impression of Change
Description: Participant-reported perception of change in impact of tinnitus on quality of life since receiving each intervention
Time Frame: 1 week post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nitrous Oxide
Number analyzed (Participants) | 37 | 37
Participants
  No change or worsened | 24 | 20
  Almost the same | 5 | 10
  A little better | 2 | 2
  Somewhat better | 4 | 0
  Moderately better | 1 | 4
  Better, definite improvement | 1 | 1
  Great deal better, considerable improvement | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 months
Groups:
- Placebo: Placebo was defined as 50% nitrogen and 50% oxygen for 40 minutes.
  Participants are blinded to the order of interventions administered. Participants have been informed prior to consent that one session will contain the nitrous oxide gas mixture, and the other session will contain the placebo gas mixture.
  Placebo gas for inhalation: Placebo gaseous mixture (50% nitrogen and 50% oxygen) for 40 minutes duration under anesthesia supervision with monitoring according to standards set by the American Society of Anesthesiologists.
- Nitrous Oxide: Nitrous oxide treatment was defined as 50% nitrous oxide and 50% oxygen for 40 minutes.
  Participants are blinded to the order of interventions administered. Participants have been informed prior to consent that one session will contain the nitrous oxide gas mixture, and the other session will contain the placebo gas mixture.
  Nitrous oxide gas for inhalation: Nitrous oxide gaseous mixture (50% nitrous oxide and 50% oxygen) for 40 minutes duration under anesthesia supervision with monitoring according to standards set by the American Society of Anesthesiologists.
Arm/Group | Placebo | Nitrous Oxide
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 3/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Nitrous Oxide (N=40)
Nausea (General disorders) | 0 (0) | 1 (1) — Temporary, fully resolved
Lightheadedness (General disorders) | 0 (0) | 1 (1) — Temporary, fully resolved
Panic attack (General disorders) | 0 (0) | 1 (1) — Temporary, fully resolved

LIMITATIONS AND CAVEATS:
Limitations included ineffective blinding, with significantly greater than 50% of participants correctly guessing the intervention received.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT03365011/Prot_SAP_000.pdf